CLINICAL TRIAL: NCT04657302
Title: A Phase I, Open-Label, Multicenter Study to Evaluate the Pharmacokinetics, Safety, Tolerability, and Efficacy of Glofitamab as Single Agent Administered After a Fixed, Single Dose Pretreatment of Obinutuzumab in Chinese Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Study to Evaluate Glofitamab as Single Agent Administered After Pretreatment With Obinutuzumab in Chinese Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YO42610
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — obinutuzumab; glofitamab; tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R/R DLBCL (Experimental): Participants will receive a fixed dose of obinutuzumab pre-treatment followed by glofitamab on Cycle 1 Days 8 and 15, then every 3 weeks (Q3W) from Cycles 2-12 (cycle length = 21 days).
  Interventions: Drug: Obinutuzumab; Drug: Glofitamab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Obinutuzumab — Participants will receive 1000 mg of intravenous (IV) obinutuzumab on Cycle 1 Day 1.
Drug: Glofitamab — Participants will receive 2.5 mg of IV glofitamab Cycle 1 Day 8, 10 mg at Cycle 1 Day 15, and 30 mg on Day 1 of Cycles 2-12 Q3W (cycle length = 21 days).
Drug: Tocilizumab — Participants will receive tocilizumab as needed to manage cytokine release syndrome (CRS).

SUMMARY:
This study will evaluate the pharmacokinetics, safety, tolerability, and efficacy of glofitamab as a single agent following a fixed single dose of obinutuzumab in Chinese patients with relapsed or refractory (R/R) diffuse large B-cell lymphoma (DLBCL) who have failed two or more lines of systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed DLBCL
* Participants must have relapsed or failed to respond to at least two lines of prior systemic therapy (including at least one prior regimen containing anthracycline, and at least one containing an anti-CD20-directed therapy)
* Participants must have measurable disease: at least one bi-dimensionally measurable nodal lesion, defined as > 1.5 cm in its longest dimension; or at least one bi-dimensionally measurable extranodal lesion, defined as > 1.0 cm in its longest dimension
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 1 or 1
* Adverse events from prior anti-cancer therapy must have resolved to Grade </=1
* Adequate liver, hematological, and renal function
* Negative serum pregnancy test within 7 days prior to study treatment in women of childbearing potential
* Women of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use contraception as defined by the protocol, and agree to refrain from donating eggs during the treatment period and for at least 18 months after the final dose of obinutuzumab, 2 months after the final dose of glofitamab, and 3 months after the final dose of tocilizumab (if applicable)
* Men must agree to remain abstinent (refrain from heterosexual intercourse) or use contraception as defined by the protocol, and agree to refrain from donating sperm during the treatment period and for at least 3 months after the final dose of obinutuzumab, 4 months after the final dose of glofitamab, and 2 months after the final dose of tocilizumab (if applicable)
* Reside in the People's Republic of China

Exclusion Criteria:

* Richter's transformation
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection within 4 weeks prior to first study treatment
* Suspected or latent tuberculosis
* Positive for HIV, hepatitis C (HCV), or hepatitis B (HBV)
* Known or suspected chronic active Epstein-Barr virus infection
* Known or suspected history of hemaphagocytic lymphohistiocytosis (HLH)
* Prior treatment with systemic immunotherapeutic agents
* History of treatment-emergent immune-related adverse events associated with prior immunotherapeutic agents
* Documented refractoriness to an obinutuzumab monotherapy-containing regimen
* Treatment with standard radiotherapy, any chemotherapeutic agent, including CAR T therapy
* Prior solid organ or allogenic stem cell transplantation
* Autologous stem cell transplantation within 100 days prior to obinutuzumab infusion
* Active autoimmune disease requiring treatment
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* History of confirmed progressive multifocal leukoencephalopathy (PML)
* Current or past history of CNS lymphoma
* Current or past history of central nervous system (CNS) disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including diabetes mellitus, history of relevant pulmonary disorders, and known autoimmune diseases
* Major surgery or significant traumatic injury < 28 days prior to obinutuzumab infusion (excluding biopsies) or anticipation of the need for major surgery during study treatment
* Another invasive malignancy in the last 2 years
* Significant cardiovascular disease
* Administration of a live, attenuated vaccine within 4 weeks before obinutizumab infusion, or anticipation that one will be required during the study
* Systemic immunosuppresive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to 3.5 years
Serum Concentration of Glofitamab | At pre-defined intervals up to 3.5 years
Total Exposure (AUC) of Glofitamab | At pre-defined intervals up to 3.5 years
Maximum Serum Concentration (Cmax) of Glofitamab | At pre-defined intervals up to 3.5 years
Minimum Serum Concentration (Cmin) of Glofitamab | At pre-defined intervals up to 3.5 years
Clearance of Glofitamab | At pre-defined intervals up to 3.5 years
Volume of Distribution at Steady State (Vss) of Glofitamab | At pre-defined intervals up to 3.5 years
Half-life (T1/2) of Glofitamab | At pre-defined intervals up to 3.5 years
Complete Response Rate (CRR) as Assessed by an Independent Review Committee (IRC) | Up to 3.5 years
Percentage of Participants with Anti-Drug Antibodies (ADA) | Up to 3.5 years

SECONDARY OUTCOMES:
Investigator-Assessed CRR | Up to 3.5 years
Objective Response Rate (ORR) as Assessed by IRC | Up to 3.5 years
ORR as Assessed by Investigator | Up to 3.5 years
Duration of Objective Response (DOR) as Assessed by IRC and Investigator | Up to 3.5 years
Duration of Complete Response (CR) as Assessed by IRC and Investigator | Up to 3.5 years
Progression-Free Survival (PFS) as Determined by IRC and Investigator | Up to 3.5 years
Overall Survival (OS) | Up to 3.5 years
Time to First Overall Response (TFOR) as Assessed by IRC and Investigator | Up to 3.5 years
Time to First Complete Response (TFCR) as Assessed by IRC and Investigator | Up to 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- China (6):
  - Beijing Cancer Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Cancer Center, Sun Yat-sen University of Medical Sciences; Department of Medical Oncology, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangsu Province Hospital, Nanjing
  - Tianjin Cancer Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).